CLINICAL TRIAL: NCT01886664
Title: Comparison of PRS According to Inhalation Agent During LDLT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Des vs Sevo PRS
Record Dates: First submitted 2012-08-20; First posted 2013-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Liver Transplantation; Postreperfusion Syndrome
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Sevoflurane (Active Comparator): Performing liver transplantation under general anesthesia using sevoflurane
  Interventions: Drug: sevoflurane
- Desflurane (Experimental): Performing liver transplantation under general anesthesia using desflurane
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: sevoflurane
  Arms: Sevoflurane
Drug: Desflurane
  Arms: Desflurane

SUMMARY:
The investigators tried to evaluate the effect of desflurane on the incidence of postreperfusion syndrome during living donor liver transplantation surgery. The investigators used sevoflurane as a comparison.

ELIGIBILITY:
Inclusion Criteria:

* elective LDLT

Exclusion Criteria:

* age < 18, age > 65
* patient refusal
* re-transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
frequency of PRS | immediately after reperfusion
  reperfusion syndrome occurs, if it occurs, immediately after reperfusion. Therefore, the primary outcome, reperfusion syndrome, can only be assessed immediately after reperfusion.

SECONDARY OUTCOMES:
ICU length of stay | after LT until the patient is transferred to the ward

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee J, Yoo YJ, Lee JM, Park YJ, Ryu HG. Sevoflurane Versus Desflurane on the Incidence of Postreperfusion Syndrome During Living Donor Liver Transplantation: A Randomized Controlled Trial. Transplantation. 2016 Mar;100(3):600-6. doi: 10.1097/TP.0000000000000874. PMID 26335917